CLINICAL TRIAL: NCT00666029
Title: Implications for Treatment of the Metabolic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2-65 (Version 4. 2007-07-03); 05/Q1704/38 (Other: Research Ethics Committee); RHM MED 0572 (Other: Southampton University Hospitals Trust R&D); 2005-000512-28 (EudraCT Number)
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Results first posted 2016-06-09 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; Volunteers recruited from the community
MeSH Terms: conditions — Metabolic Syndrome | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Active Comparator): Active arm atorvastatin 40 mg. o.d.
  Interventions: Drug: atorvastatin
- Placebo (Placebo Comparator): Placebo arm dummy pill
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: atorvastatin — 40 m.g. o.d. tablets for 6 months
  Other Names: Lipitor
  Arms: Atorvastatin
Drug: placebo — Placebo
  Other Names: Dummy
  Arms: Placebo

SUMMARY:
To characterize features of metabolic syndrome in volunteers. To undertake a randomised trial to determine whether treatment with a statin improves muscle microvascular blood flow.

DETAILED DESCRIPTION:
To characterise features of the metabolic syndrome, including body fat, insulin sensitivity, and liver fat together with muscle micorvascular blood flow.

To undertake a randomised controlled trial of atorvastatin 40 mg. o.d for 6 months to determine whether any of the above measures change with treatment.

ELIGIBILITY:
Inclusion criteria Body mass index (BMI) 20-35 kg/m^2" and "> 3 criteria for the metabolic syndrome (NCEP III ATP criteria - see below) , one of which will be hypertriglyceridaemia, i.e. fasting plasma triglycerides >2.0 mmol/L - a cardinal lipid abnormality of the syndrome

NCEP III ATP metabolic syndrome criteria are:

Waist greater than or equal to 102 cm BP greater than 130 / 85 mmHg TG greater than or equal to 1.7mmol/l Glucose greater than or equal to 6.1 mmol/l HDL less than 1.0 mmol/l

Exclusion Criteria:

Aged <18 years Aged >75 years Known diabetes; renal, liver, or uncontrolled thyroid disease; uncontrolled hypertension; treatment with lipid-modifying drugs; antihypertensive medication; corticosteroid therapy; or hormone replacement therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Clough GF, Turzyniecka M, Walter L, Krentz AJ, Wild SH, Chipperfield AJ, Gamble J, Byrne CD. Muscle microvascular dysfunction in central obesity is related to muscle insulin insensitivity but is not reversed by high-dose statin treatment. Diabetes. 2009 May;58(5):1185-91. doi: 10.2337/db08-1688. Epub 2009 Feb 10. PMID 19208914
- [Result] Turzyniecka M, Wild SH, Krentz AJ, Chipperfield AJ, Gamble J, Clough GF, Byrne CD. Skeletal muscle microvascular exchange capacity is associated with hyperglycaemia in subjects with central obesity. Diabet Med. 2009 Nov;26(11):1112-9. doi: 10.1111/j.1464-5491.2009.02822.x. PMID 19929989
- [Result] Turzyniecka M, Wild SH, Krentz AJ, Chipperfield AJ, Clough GF, Byrne CD. Diastolic function is strongly and independently associated with cardiorespiratory fitness in central obesity. J Appl Physiol (1985). 2010 Jun;108(6):1568-74. doi: 10.1152/japplphysiol.00023.2010. Epub 2010 Mar 25. PMID 20339006
- [Result] Clough GF, L'Esperance V, Turzyniecka M, Walter L, Chipperfield AJ, Gamble J, Krentz AJ, Byrne CD. Functional dilator capacity is independently associated with insulin sensitivity and age in central obesity and is not improved by high dose statin treatment. Microcirculation. 2011 Jan;18(1):74-84. doi: 10.1111/j.1549-8719.2010.00070.x. PMID 21166928

RESULTS

PARTICIPANT FLOW:
Groups:
- Atorvastatin: Active arm atorvastatin 40 mg. o.d.
  Participants randomised to atorvastatin: 40 m.g. o.d. tablets for 6 months
Period: Overall Study
Arm/Group | Atorvastatin | Placebo
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Age 18-75 years, body mass index (BMI) 20-35 kg/m2, with > 3 criteria for the metabolic syndrome.
  (One person in the placebo arm did not have complete baseline data).
Groups:
- Atorvastatin: Active arm atorvastatin 40 mg. o.d.
  atorvastatin: 40 m.g. o.d. tablets for 6 months Age 18-75 years, body mass index (BMI) 20-35 kg/m2, with > 3 criteria for the metabolic syndrome , one of which will be hypertriglyceridaemia, i.e. fasting plasma triglycerides >2.0 mmol/L - a cardinal lipid abnormality of the syndrome.
- Placebo: Placebo arm dummy pill
  placebo: Placebo Age 18-75 years, body mass index (BMI) 20-35 kg/m2, with > 3 criteria for the metabolic syndrome , one of which will be hypertriglyceridaemia, i.e. fasting plasma triglycerides >2.0 mmol/L - a cardinal lipid abnormality of the syndrome.
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Placebo | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 39
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (9.0) | 51.4 (9.0) | 51.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Muscle Microvascular Function
Description: Skeletal muscle microvascular function assessed (Filtrass plethysmographic system) using a passive inductive transducer (Compumedics.dwl, Singen, Germany) and a small pressure step venous congestion protocol. Fluid filtration rate (Jv mL min-1 100 mL-1), measured from the slope of limb volume change in response to each pressure step (10 mmHg steps to 60 mmHg around the thigh) over the last 2 minutes of its application, to allow for completion of vascular filling, and plotted against cuff pressure (Pcuff). The slope of this relationship, at pressures above those giving rise to net filtration, is a measure of Kf, microvascular filtration capacity, a function of exchange surface area and permeability. The CV for Kf measurement was 14.5%.
Time Frame: 6 months
Population: There was missing data on two participants in the atorvastatin arm and two participants in the placebo arm.
Measure: Mean (Standard Deviation); unit: 10^3 mL*min^-1*100ml^-1*mmHg^-1
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 17 | 18
10^3 mL*min^-1*100ml^-1*mmHg^-1 | 3.7 (1.4) | 4.0 (1.1)

2. Primary Outcome: Insulin Sensitivity Index
Description: Insulin sensitivity index was assessed during the final steady state 30 minutes of a high dose hyperinsulinaemic euglycaemic clamp (insulin infusion rate 1.5 mIU/kg/min). During this part of the clamp, insulin was infused at 1.5mIU/kg/min and the glucose concentration was maintained at 5 mmol/L using a dextrose infusion. The whole body insulin mediated glucose disposal rate (M value - mg/kg/min) was estimated from the total amount of glucose infused during the last 30 minutes of the clamp. The mean of four serum insulin concentrations was taken during this 30 minutes to determine the steady state insulin concentration (I value - milliunits/litre). M value/I value defined the insulin sensitivity index.
Time Frame: 6 months
Population: There was missing data in four people in the atorvastatin arm and two people in the placebo arm
Measure: Mean (Standard Deviation); unit: mg*kg^-1*min^-1*mIU^-1*L^-1
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 15 | 18
mg*kg^-1*min^-1*mIU^-1*L^-1 | 0.56 (0.21) | 0.41 (0.14)

ADVERSE EVENTS:
Time Frame: Adverse event data collected over 6 months
Arm/Group | Atorvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (N=20) | Placebo (N=20)
muscle ache (Musculoskeletal and connective tissue disorders) | 1 | 0 — Muscle ache on medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes